CLINICAL TRIAL: NCT05751629
Title: Cohort A: PARP Inhibitor-Naïve Platinum-Resistant Ovarian Cancer Treatment Cohort With TSR-042, Bevacizumab, and Niraparib
Brief Title: Study to Evaluate the Safety and Efficacy of TSR-042, Bevacizumab, and Niraparib in Participants With Recurrent Ovarian Cancer
Acronym: COHORT-A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 213357-COHORT-A
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-02

CONDITIONS: Ovarian Neoplasm
Keywords: Poly-ADP-ribose polymerase (PARP) Inhibitor; Ovarian cancer; Niraparib; Bevacizumab; TSR-042; Neoadjuvant treatment
MeSH Terms: conditions — Ovarian Neoplasms | interventions — dostarlimab; Bevacizumab; niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort A (Dostarlimab + Bevacizumab + Niraparib) (Experimental)
  Interventions: Drug: Dostarlimab; Drug: Bevacizumab; Drug: Niraparib

INTERVENTIONS:
Drug: Dostarlimab — Dostarlimab was administered.
  Other Names: TSR-042
Drug: Bevacizumab — Bevacizumab was administered.
  Other Names: Avastin
Drug: Niraparib — Niraparib was administered.
  Other Names: ZEJULA

SUMMARY:
The primary objective of this sub study is to evaluate the efficacy of the combination of TSR-042, bevacizumab, and niraparib in participants with advanced, relapsed, high-grade ovarian, fallopian tube, or primary peritoneal cancer who have received 1 to 2 prior lines of anticancer therapy, are PARP inhibitor naïve, and have platinum-resistant but not refractory disease.

This study is a sub study of the master protocol - OPAL (NCT03574779).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be resistant to the most recent platinum-based therapy, defined for the purpose of this protocol as progression within 6 months from completion of a minimum of 4 cycles of platinum-containing therapy. This should be calculated from the date of the last administered dose of platinum therapy to the date of the radiographic imaging showing disease progression. Participant with primary platinum-refractory disease as defined by those who progressed during or within 4 weeks of completion of first platinum-based chemotherapy are not eligible
* Participant must not have received any prior therapy for ovarian cancer with a PARP inhibitor
* Participant has had 1 to 2 prior lines of anticancer therapy for ovarian cancer
* Participant is able to take oral medications.

Exclusion Criteria:

* Participant has known hypersensitivity to TSR-042, bevacizumab, niraparib, their components, or their excipients
* Participant has a known history of myelodysplastic syndrome or acute myeloid leukemia
* Participant has active autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* Participant received prior treatment with an anti- programmed death-1 (PD-1) or anti- programmed death-ligand 1 (PD-L1) agent
* Participant has received prior treatment with anti-angiogenic therapy with the exception of bevacizumab. (Participant who received prior bevacizumab are eligible only if they did not discontinue bevacizumab due to toxicity, as established by the Investigator.)
* Participant has bowel obstruction, had bowel obstruction within the past 3 months, or is otherwise judged by the Investigator to be at high risk for bowel obstruction related to the underlying disease. Participant has any history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscesses. Evidence of recto-sigmoid involvement by pelvic examination or significant bowel involvement on computed tomography scan
* Participant has proteinuria as demonstrated by urine protein:creatinine ratio ≥1.0 at screening or urine dipstick for proteinuria ≥2 (Participant discovered to have ≥2 proteinuria on dipstick at baseline should undergo 24-hour urine collection and must demonstrate <2g of protein in 24 hours to be eligible.)
* Participant is at increased bleeding risk due to concurrent conditions (eg, major injuries or surgery within the past 28 days prior to start of study treatment, history of hemorrhagic stroke, transient ischemic attack, subarachnoid hemorrhage, or clinically significant hemorrhage within the past 3 months)
* Participant has a history of recent major thromboembolic event defined as follows:

  1. Pulmonary embolism diagnosed within 3 months of enrollment
  2. Lower extremity deep venous thrombosis diagnosed within 3 months of enrollment (Participant with a history of thromboembolic disease on stable therapeutic anticoagulation for more than 3 months prior to enrollment are eligible for this study.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female participants will be included.
Enrollment: 41 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- United States (9):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Palo Alto, California
  - GSK Investigational Site, Ventura, California
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: http://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study is a sub study of the master protocol (NCT03574779).
Groups:
- Cohort A (Dostarlimab + Bevacizumab + Niraparib): Participants with platinum-resistant advanced, relapsed, high-grade ovarian, fallopian tube, or primary peritoneal cancer, and poly(adenosine diphosphate [ADP] ribose) polymerase [PARP] inhibitor naive were administered 500 milligrams (mg) of Dostarlimab (TSR-042) via infusion on Day 1 every 3 weeks (Q3W) for 4 cycles (each cycle is of 21 days), followed by 1000 mg every 6 weeks (Q6W) beginning from Day 1 of Cycle 5 until progressive disease (PD) or toxicity. Participants were administered 15 milligram per kilogram (mg/kg) of Bevacizumab via infusion Q3W for up to 15 months. Participants with screening actual body weight greater than or equal (≥) to 77 kg and screening platelet count ≥ 150000 cells per microliter were administered 300 mg of Niraparib orally once daily throughout each 21-day cycle until PD or toxicity. Participants with screening actual body weight less than 77 kg or screening platelet count less than 150000 cells per microliter were administered 200 mg of niraparib orally, once daily throughout each 21-day cycle until PD or toxicity.
Period: Overall Study
Arm/Group | Cohort A (Dostarlimab + Bevacizumab + Niraparib)
Started | 41
Completed | 0
Not Completed | 41
Not completed — Withdrawal by Subject | 6
Not completed — Death | 25
Not completed — Study Site Closed | 9
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cohort A (Dostarlimab + Bevacizumab + Niraparib)
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (10.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 32
  More than one race | 0
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 by Investigator Assessment
Description: ORR was defined as percentage of participants with a confirmed investigator-assessed Best Overall Response (BOR) of confirmed complete response (CR) or partial response (PR), evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. CR is defined as the disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm).
Time Frame: Up to approximately 38 Months
Population: Response-evaluable population included all efficacy participants (all participants who received any amount of study treatment with measurable disease at baseline) with at least 1 evaluable post-baseline tumor assessment.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A (Dostarlimab + Bevacizumab + Niraparib)
Number analyzed (Participants) | 39
Percentage of participants | 17.9 [10.3 to 28.3]

2. Secondary Outcome: Progression Free Survival (PFS) Per RECIST Version 1.1 by Investigator Assessment
Description: PFS was defined as the time from the date of the first dose of study treatment to the earliest date of assessment of disease progression or death by any cause in the absence of progression by RECIST v1.1. Disease Progression is defined using RECIST v1.1 as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to approximately 38 Months
Population: Efficacy Population included all safety participants (all participants who received any amount of study treatment) with measurable disease at baseline. Measurable disease at baseline was defined by the existence of at least 1 target lesion at baseline tumor assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A (Dostarlimab + Bevacizumab + Niraparib)
Number analyzed (Participants) | 41
Months | 7.92 [4.17 to 10.87]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of the first dose of study treatment to the date of death due to any cause. Median and 95% CI are presented.
Time Frame: Up to approximately 38 Months
Population: Efficacy Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A (Dostarlimab + Bevacizumab + Niraparib)
Number analyzed (Participants) | 41
Months | 22.05 [11.14 to 26.25]

4. Secondary Outcome: Duration of Response (DOR) Per RECIST Version 1.1 by Investigator Assessment
Description: DOR was defined as the time from first documentation of response (CR or PR) until the time of first documentation of disease progression by RECIST version 1.1 based on Investigator's assessment or death by any cause. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm).
Time Frame: Up to approximately 38 Months
Population: Response-evaluable population. Only responders by investigator were included in this analysis.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cohort A (Dostarlimab + Bevacizumab + Niraparib)
Number analyzed (Participants) | 11
Months | 11.76 [4.86 to 23.98]

5. Secondary Outcome: Disease Control Rate (DCR) Per RECIST Version 1.1 by Investigator Assessment
Description: DCR was defined as the percentage of participants who have achieved best overall response of CR, PR, or stable disease (SD) per RECIST version 1.1 based on Investigator's assessment. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm). Stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Up to approximately 38 Months
Population: Response-evaluable population.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A (Dostarlimab + Bevacizumab + Niraparib)
Number analyzed (Participants) | 39
Percentage of participants | 76.9 [66.0 to 85.6]

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Time Frame: Up to approximately 38 Months
Population: Safety population included all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Dostarlimab + Bevacizumab + Niraparib)
Number analyzed (Participants) | 41
Participants | 41

7. Secondary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Parameters - Chemistry, Coagulation, Hematology and Thyroid
Description: Blood samples were collected for the analysis of clinical laboratory parameters - chemistry, coagulation, hematology and thyroid.
Time Frame: Up to approximately 38 Months
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Dostarlimab + Bevacizumab + Niraparib)
Number analyzed (Participants) | 41
Participants | 0

8. Secondary Outcome: Absolute Values in Urinalysis Parameter - Specific Gravity (Ratio)
Description: Urine samples were collected at indicated time points for the assessment of specific gravity. Baseline is defined as the most recent non-missing measurement prior to or on the first administration of study drug.
Time Frame: Baseline (Day 1) and end of treatment (Up to approximately 32 months)
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort A (Dostarlimab + Bevacizumab + Niraparib)
Number analyzed (Participants) | 36
Ratio
  Baseline | 1.0149 (0.00794)
  End of treatment: number analyzed (Participants) | 26
  End of treatment | 1.0162 (0.00786)

9. Secondary Outcome: Change From Baseline in Cancer Antigen 125 (CA-125) at End of Treatment
Description: Blood samples were collected for the analysis of CA-125. Baseline is defined as the most recent non-missing measurement prior to or on the first administration of study drug.
Time Frame: Baseline (Day 1) and end of treatment (Up to approximately 32 months)
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per milliliter (U/mL)
Arm/Group | Cohort A (Dostarlimab + Bevacizumab + Niraparib)
Number analyzed (Participants) | 37
Units per milliliter (U/mL) | 246.86 (608.985)

10. Secondary Outcome: Change From Baseline in Vital Signs (Weight) at End of Treatment
Description: Weight was measured in ordinary indoor clothing (without shoes) and was recorded at specified study visit. Baseline is defined as the most recent non-missing measurement prior to or on the first administration of study drug.
Time Frame: Baseline (Day 1) and end of treatment (Up to approximately 32 months)
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Cohort A (Dostarlimab + Bevacizumab + Niraparib)
Number analyzed (Participants) | 36
kilogram | -5.07 (5.475)

11. Secondary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status at Baseline and End of Treatment
Description: Performance status assessments were based on 5-grade ECOG scale (from 0 to 4), where 0=fully active, able to carry on all pre-disease performance without restriction; 1=restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (e.g., light house work, office work); 2=ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours; 3=capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4=completely disabled, cannot carry on any self-care, totally confined to bed or chair. Baseline is defined as the most recent non-missing measurement prior to or on the first administration of study drug.
Time Frame: Baseline (Day 1) and end of treatment (Up to approximately 32 months)
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Dostarlimab + Bevacizumab + Niraparib)
Number analyzed (Participants) | 40
Participants
  Baseline: Grade 0 | 18
  Baseline: Grade 1 | 22
  Baseline: Grade 2 | 0
  Baseline: Grade 3 | 0
  Baseline: Grade 4 | 0
  End of Treatment: number analyzed (Participants) | 37
  End of Treatment: Grade 0 | 9
  End of Treatment: Grade 1 | 20
  End of Treatment: Grade 2 | 7
  End of Treatment: Grade 3 | 1
  End of Treatment: Grade 4 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious advents (Non-SAEs) and serious adverse events (SAE) were collected up to 38 months.
Description: Safety population included all participants who received any amount of study treatment.
Arm/Group | Cohort A (Dostarlimab + Bevacizumab + Niraparib)
All-Cause Mortality (participants affected / at risk) | 25/41
Serious Adverse Events (participants affected / at risk) | 22/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (Dostarlimab + Bevacizumab + Niraparib) (N=41)
Small intestinal obstruction (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
COVID-19 (Infections and infestations) | 1
Human anaplasmosis (Infections and infestations) | 1
Parainfluenzae virus infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Viral rash (Infections and infestations) | 1
Vulval abscess (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Immune-mediated cytopenia (Blood and lymphatic system disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Chest pain (General disorders) | 1
Pyrexia (General disorders) | 1
Seizure (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Dostarlimab + Bevacizumab + Niraparib) (N=41)
Nausea (Gastrointestinal disorders) | 28 (47)
Vomiting (Gastrointestinal disorders) | 23 (47)
Abdominal pain (Gastrointestinal disorders) | 16 (22)
Constipation (Gastrointestinal disorders) | 15 (27)
Diarrhoea (Gastrointestinal disorders) | 14 (19)
Abdominal distension (Gastrointestinal disorders) | 8 (9)
Stomatitis (Gastrointestinal disorders) | 5 (10)
Abdominal discomfort (Gastrointestinal disorders) | 4 (5)
Ascites (Gastrointestinal disorders) | 4 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (4)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (4)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 2 (3)
Haemorrhoids (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 2 (2)
Anal incontinence (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (2)
Dental caries (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (2)
Gingival bleeding (Gastrointestinal disorders) | 1 (2)
Gingival ulceration (Gastrointestinal disorders) | 1 (2)
Oral disorder (Gastrointestinal disorders) | 1 (1)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (3)
Oral pruritus (Gastrointestinal disorders) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1)
Short-bowel syndrome (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 17 (51)
Aspartate aminotransferase increased (Investigations) | 15 (24)
Blood creatinine increased (Investigations) | 11 (17)
Neutrophil count decreased (Investigations) | 11 (29)
Alanine aminotransferase increased (Investigations) | 10 (27)
Blood alkaline phosphatase increased (Investigations) | 9 (17)
Weight decreased (Investigations) | 7 (9)
Amylase increased (Investigations) | 4 (4)
Blood chloride decreased (Investigations) | 4 (4)
Blood lactate dehydrogenase increased (Investigations) | 4 (5)
White blood cell count decreased (Investigations) | 4 (21)
Blood thyroid stimulating hormone increased (Investigations) | 3 (6)
Lymphocyte count decreased (Investigations) | 3 (5)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
International normalised ratio increased (Investigations) | 2 (4)
Blood albumin increased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Blood urea increased (Investigations) | 1 (2)
Carbohydrate antigen 125 increased (Investigations) | 1 (1)
Neutrophil count increased (Investigations) | 1 (1)
Protein total decreased (Investigations) | 1 (1)
Protein total increased (Investigations) | 1 (2)
Prothrombin time prolonged (Investigations) | 1 (1)
Thyroxine free increased (Investigations) | 1 (1)
Troponin increased (Investigations) | 1 (2)
Urine protein/creatinine ration increased (Investigations) | 1 (2)
Fatigue (General disorders) | 30 (59)
Pyrexia (General disorders) | 8 (18)
Oedema peripheral (General disorders) | 7 (8)
Mucosal inflamation (General disorders) | 4 (4)
Chest pain (General disorders) | 3 (4)
Malaise (General disorders) | 3 (3)
Asthenia (General disorders) | 1 (1)
Catheter site pruritus (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Ulcer (General disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 15 (24)
Hyponatraemia (Metabolism and nutrition disorders) | 14 (22)
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 (11)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (12)
Hypernatraemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (22)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (16)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (12)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (9)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 19 (69)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (16)
Lymphopenia (Blood and lymphatic system disorders) | 5 (23)
Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (10)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 10 (19)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 2 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 20 (41)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Flushing (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Headache (Nervous system disorders) | 16 (23)
Dizziness (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 3 (3)
Taste disorder (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Disturbance in attention (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (2)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5)
Sinusitis (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Abdominal abcess (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Catheter site cellulitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Lyme disease (Infections and infestations) | 1 (2)
Oesophageal candidiasis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Viral rash (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 14 (21)
Anxiety (Psychiatric disorders) | 4 (4)
Nervousness (Psychiatric disorders) | 1 (2)
Sleep disorder (Psychiatric disorders) | 1 (2)
Proteinuria (Renal and urinary disorders) | 8 (18)
Pollakiuria (Renal and urinary disorders) | 4 (4)
Dysuria (Renal and urinary disorders) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (2)
Post procedural contusion (Injury, poisoning and procedural complications) | 1 (1)
Hypothyroidism (Endocrine disorders) | 7 (10)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Palpitations (Cardiac disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (2)
Tachycardia (Cardiac disorders) | 1 (3)
Vision blurred (Eye disorders) | 3 (4)
Cataract (Eye disorders) | 2 (2)
Eye pruritus (Eye disorders) | 1 (1)
Eye swelling (Eye disorders) | 1 (1)
Macular degeneration (Eye disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 2 (2)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 (1)
Genital rash (Reproductive system and breast disorders) | 1 (1)
Pelvic discomfort (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1)
Inner ear disorder (Ear and labyrinth disorders) | 1 (2)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Multiple allergies (Immune system disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Abdominal cavity drainage (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT05751629/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT05751629/SAP_001.pdf